CLINICAL TRIAL: NCT05743777
Title: A Phase II Study of PembROlizumab With or Without Microbial EcOsystem ThErapeutic 4 (MET4) in Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: PembROlizumab With or Without Microbial EcOsystem ThErapeutic 4 (MET4) in Advanced Head and Neck Squamous Cell Carcinoma
Acronym: PROMOTE-HN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company withdrew financial support
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HN12
Record Dates: First submitted 2023-02-09; First posted 2023-02-24 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + MET-4 (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: MET-4
- Pembrolizumab + Placebo (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — 400 mg IV q6 weekly for a maximum of 18 cycles
Drug: MET-4 — Cycle 1: 5 g (10 capsules) on days -7 and -6 and 1.5 g (3 capsules) on day -5 and every day thereafter Cycle 2 onwards: 1.5 g (3 capsules) daily
  Arms: Pembrolizumab + MET-4
Drug: Placebo — Cycle 1: 5 g (10 capsules) on days -7 and -6 and 1.5 g (3 capsules) on day -5 and every day thereafter Cycle 2 onwards: 1.5 g (3 capsules) daily
  Arms: Pembrolizumab + Placebo

SUMMARY:
The usual approach for patients who are not in a study is treatment with pembrolizumab, a type of immunotherapy drug. Immunotherapy works by allowing the immune system to detect your cancer and reactivate the immune response. This may help to slow down the growth of cancer and may cause cancer cells to die.

DETAILED DESCRIPTION:
This study is being done to answer the following question: Can the addition of a new treatment improve the cancer-shrinking ability of the usual treatment in patients with advanced head and neck cancer?

This study is being done in order to find out if this approach is better or worse than the usual approach for advanced head and neck cancer. The usual approach is defined as the care most people get for advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically-confirmed R/M HNSCC considered incurable by local therapies.
* Patients must not have had any prior systemic therapy administered in the recurrent or metastatic setting.
* Patients with prior systemic therapy given as part of multimodal treatment for locoregionally advanced disease must have completed treatment > 6 months prior to signing consent.
* Patients must have one of the following primary tumor locations: oropharynx, oral cavity, hypopharynx, and larynx. Primary tumor site of nasopharynx (any histology) is excluded.
* Patients with oropharyngeal cancer, must have Human Papilloma Virus (HPV) status determined by p16 immunohistochemical staining on a tumor specimen. Local testing is acceptable.
* Patients must be at least 18 years of age on day of signing informed consent.
* Patients must have measurable disease based on RECIST 1.1 as determined by the site. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Patients must have an ECOG performance status of 0 or 1
* Abs neutrophil count ≥1,500/μL; Platelets ≥ 100,000; Hemoglobin ≥9 g/dL; Creatinine or measured or calculated creatinine clearance ≤ 1.5 x UNL or ≥ 30mL/min for subject with creatinine levels > 1.5 x UNL; Total bilirubin ≤ 1.5 x UNL or Direct bilirubin ≤ UNL for subjects with total bilirubin levels > 1.5 x ULN; ALT ≤ 2.5 UNL or ≤ 5 x UNL for subjects with liver metastases
* Patients must have PD-L1 positive (CPS ≥1) tumor as determined by PD-L1 testing performed at the local laboratory, from a core or excisional biopsy (fine needle aspirate is not adequate).
* Patients must consent to provision of samples of blood, oropharyngeal swab, and stool for correlative marker analysis.
* Patients must consent to the submission of, and investigator must confirm access to and agree to submit within 4 weeks of enrollment, a formalin-fixed, paraffin-embedded tumour (FFPE) tissue block, cores (two 2 mm cores of tumour from the block), or 10-15 freshly cut unstained tumour slides (4 µm thick) for protocol-mandated exploratory assessments.
* Patient must be able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French
* Women of childbearing potential must have a negative blood pregnancy test within 72 hours prior to receiving the first dose of study medication to confirm eligibility as part of the Pre-Study Evaluation
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method starting with first dose of study therapy through 180 days after the last dose of study therapy
* Patients must be able to swallow oral medications.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrolment in the trial to document their willingness to participate.

Exclusion Criteria:

* Patients with disease that is suitable for local therapy administered with curative intent.
* Patients with progressive disease (PD) within six (6) months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.
* Patients with persisting toxicity related to prior therapy Grade >2 constituting a safety risk based on the investigator's judgement.
* Patients with a history of a gastrointestinal condition or procedure that, in the opinion of the investigator, may affect oral study drug absorption.
* Patients currently participating and receiving study therapy, or that have participated in a study of an investigational agent and received study therapy, or used an investigational device, any of which occurred within 4 weeks of the first dose of treatment.
* Patients with life expectancy of less than 3 months and/or that have rapidly progressing disease (e.g. tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
* Patients with diagnosis of immunodeficiency or that are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Corticosteroid use as pre-medication for allergic reactions (e.g. IV contrast) is allowed. The use of physiologic doses of corticosteroids (e.g.: prednisone ≤10 mg/days) is allowed.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 3 years. Other exceptions may be considered with CCTG consultation.
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patients with active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Patients with allogeneic tissue/solid organ transplant.
* Patients with active infection requiring systemic therapy.
* Patients that have had prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent or any other immune compounds.
* Patients with known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Subjects with well controlled Human Immunodeficiency Virus (HIV) are allowed.
* Patients that have received live vaccine within 30 days of planned start of study therapy. COVID19 vaccination will be allowed and should be recorded as concomitant medication.
* Patients with history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Patients that are pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate per RECIST 1.1 in first line recurrent and/or metastatic (R/M) HNSCC subjects, treated with pembrolizumab in combination with MET-4 or pembrolizumab with placebo. | 3 years

SECONDARY OUTCOMES:
Progression-free survival as per RECIST 1.1 | 3 years
Overall survival | 3 years
Duration of response | 3 years
Number and severity of adverse events per CTCAE version 5.0 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, Study Chair — University Health Network, Princess Margaret Cancer Centre, Toronto ON Canada

IPD SHARING:
Plan to Share IPD: No